CLINICAL TRIAL: NCT06997081
Title: Elranatamab, Lenalidomide, Dexamethasone in Newly Diagnosed Multiple Myeloma, a Clinical and Correlative Phase 2 Study
Brief Title: ERd Combination Treatment in Newly Diagnosed Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Carl Ola Landgren, MD, PhD, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20250076
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Elranatamab in combination with lenalidomide and dexamethasone (ERd) (Experimental): Participants in this group will receive standard of care (SOC) therapy with ERd combination treatment.
  Total participation duration is up to 2.5 years.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Drug: Elranatamab

INTERVENTIONS:
Drug: Lenalidomide — Participants will receive 25mg of Lenalidomide orally on Days 2-21 of Cycle 1, then 25 mg by mouth on Days 1-21 of the remaining cycles.
Drug: Dexamethasone — Participants will receive 20mg of Dexamethasone orally on Days 1, 3, 8, and 15 of Cycle 1, then 4mg orally on Days 1 and 15 of Cycles 4-6.
Drug: Elranatamab — Participants will receive 12mg Elranatamab subcutaneous (SC) on Cycle 1; 32mg subcutaneous (SC) on Cycle 1 Day 3; 76mg subcutaneous (SC) on Cycle 1 Day 8 and Day 15. Then, participants will receive 76mg subcutaneous (SC) on Days 1 and 15 of Cycles 2-6. Lastly, participants will receive Elranatamab subcutaneous (SC) on Day 1 of the remaining cycles.

SUMMARY:
The purpose of this study is to determine the effects that Elranatamab in combination with Lenalidomide and Dexamethasone has on participants that have been newly diagnosed with Multiple Myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed patients with histologically confirmed multiple myeloma (MM) based on the IMWG diagnostic criteria and measurable disease within the past 4 weeks (or past 8 weeks if patient received pre-study MM therapy) based on one of the following:

   * Serum monoclonal protein ≥ 1.0 g/dL
   * Urine monoclonal protein ≥ 200 mg/24 hour
   * Involved serum immunoglobulin free light chain ≥ 10 mg/dL AND abnormal kappa/lambda ratio

   Note:
   * Patients who have evaluable disease based on samples other than urine do not need to have urine evaluated for initial or subsequent response assessments.
   * Because the primary endpoint is MRD negativity rate, per the discretion of the Principal Investigator (PI), patients without measurable disease (e.g., M-spike <1.0 g/dL) may also be enrolled in line with the International Myeloma Working Group (IMWG) MM response criteria.
2. Evidence of underlying end organ damage and/or myeloma defining event attributed to underlying plasma cell proliferative disorder meeting at least one of the following (Note: Myeloma defining event does not need to be based on repeat testing done at screening if previous pathology, radiology, etc., confirm diagnosis of myeloma per IMWG):

   * Hypercalcemia: serum calcium >0.25 mmol/L (>1.0 mg/dL) above upper limit of normal (ULN) or ≥2.75 mmol/L (11 mg/dL)
   * Anemia: hemoglobin value <10 g/dL or >2 g/dL below lower limit of normal (LLN)
   * Bone disease: ≥1 lytic lesions on skeletal X-ray, computed tomography (CT), or positron emission tomography (PET)-CT. For patients with 1 lytic lesion, bone marrow should demonstrate ≥10% clonal plasma cells
   * Clonal bone marrow plasma cell percentage ≥60%
   * Involved/un-involved serum free light chain ratio ≥100 and involved free light chain ≥100 mg/L.
   * >1 focal lesion on magnetic resonance imaging study (lesion must be >5 mm) in size
   * For patients with 1 lytic lesion, bone marrow should demonstrate ≥10% clonal plasma cells
3. Patients must have measurable disease within the past 4 weeks, which is defined by any one of the following:

   * Serum monoclonal protein ≥ 0.5 g/dL Urine monoclonal protein >200 mg/24 hour
   * Serum immunoglobulin free light chain ≥10 mg/dL AND abnormal kappa/lambda serum free light chain ratio (reference: 0.26-1.65)
   * Other measurable disease as defined by the IMWG
   * Because the primary endpoint is MRD negativity based on bone marrow analysis, a patient without measurable disease in blood or urine may be enrolled and assessed for MRD negativity.

   Note:
   * Participants who have evaluable disease based on samples other than urine do not need to have urine evaluated for subsequent responses.
   * In participants who received minimal prior therapy within the allowable range per exclusion criteria 1, patients should have had documented measurable disease within 4 weeks of starting that respective therapy if currently unmeasurable.
4. Adult male and female participants ≥ 18 years of age.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Refer to Appendix A)
6. Participants must have adequate organ and marrow function ≤45 days as defined below:

   * Absolute neutrophil count (ANC) >1.0 K cells/μL; At the discretion of the Investigator, patients with an ANC of 0.5 K/μL-1.0 K/μL may also be enrolled if clinically appropriate (eg, patients with a baseline neutropenia that is chronic and/or ethnic neutropenia and that does not cause complications, e.g, no history of chronic infections).
   * Platelet count >75 K cells/μL
   * Hemoglobin >8 g/dL (transfusions are permissible if the cause of the anemia is other than myeloma)
   * Total bilirubin <1.5 X upper limit of normal (ULN).
   * Note: Isolated total bilirubin ≥1.5 X ULN with conjugated [direct] bilirubin <1.5 X ULN is allowed for those participants with known Gilbert's syndrome.
   * Aspartate aminotransferase (AST)/ alanine transaminase (ALT) ≤2.5 X ULN
   * GFR ≥30 mL/min based on Modification of Diet in Renal Disease (MDRD) 4-variable Formula calculation (Appendix 17.2) or creatine clearance (CrCl) measured by a 24-hour urine collection. (The estimated glomerular filtration rate (eGFR) may also be determined by using other widely accepted methods as clinically indicated, ie, Cockcroft-Gault method or the chronic kidney disease (CKD)-epidemiology collaboration (EPI) per institutional standards.
7. Participants must be willing, able, and agree to enrolling in the lenalidomide Risk Evaluation and Mitigation Strategy (REMS) program.
8. A female participant of childbearing potential must have a negative serum or urine pregnancy test at screening (at or within 45 days of study enrollment) and within 72 hours of the start of study treatment and must agree to further serum or urine pregnancy tests during the study
9. A female participant must be:

   * Not of childbearing potential, or
   * Of childbearing potential and practicing at least 1 highly effective method of contraception as described in Section 5.7
10. A female participant must agree not to donate eggs (ova, oocytes) or freeze for future use for the purposes of assisted reproduction during the study and for at least 4 weeks after the last dose of lenalidomide or 4 months after the last dose of elranatamab. Female participants should consider preservation of eggs prior to study treatment, as anti-cancer treatments may impair fertility.
11. A female participant must agree to not breastfeed during the study and for a period of at least 4 weeks after the last dose of lenalidomide or 4 months after the last dose of elranatamab.
12. A male participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person during the study and for a period of at least 4 weeks after receiving the last dose of study treatment. If the male participant's partner is a female of childbearing potential, the male participant must use condoms (with or without spermicide), and the female partner of the male participant must also be practicing a highly effective method of contraception. Refer to Section 5.7 for contraception requirements.

    Note: If the male participant is vasectomized, he still must wear a condom (with or without spermicidal foam/gel/film/cream/suppository), but his female partner is not required to use contraception.
13. A male participant must agree not to donate sperm for the purpose of reproduction during the study and for period of 3 months after receiving the last dose of study treatment. Male participants should consider preservation of sperm prior to study treatment, as anti-cancer treatments may impair fertility.
14. Ability of the patient to understand and the willingness to sign a written informed consent document.
15. Have any condition that, in the opinion of the Investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements.
16. Must be willing and able to adhere to the lifestyle restrictions specified in this protocol.

Exclusion Criteria:

1. Participants receiving >1 cycle of prior treatment or concurrent systemic treatment for MM with the following exceptions:

   * Treatment of hypercalcemia or spinal cord compression or aggressively progressing myeloma with current or prior corticosteroids is permitted
   * Bone targeting agents are permitted
   * Concurrent or prior treatment with corticosteroids for indications other than multiple myeloma is permitted
   * Prior MM treatments, such as immunomodulatory drugs (IMIDs) or non-MM drugs in clinical trials for smoldering myeloma is permitted with a washout period of 2 weeks from last dose. Patients with Smoldering Multiple Myeloma (SMM) previously treated with carfilzomib are excluded.
   * Patients with measurable disease who received up to one cycle of any therapy within 60 days with a washout period of 2 weeks from last dose (on a trial or outside a trial) are eligible (Note: Measurable disease is defined as one or more of the following: Serum monoclonal protein ≥ 1.0 g/dL, Urine monoclonal protein ≥ 200 mg/24 hour and/or involved serum immunoglobulin free light chain ≥ 10 mg/dL AND abnormal kappa/lambda ratio.)
2. Known active central nervous system (CNS) involvement or clinical signs of myelomatous meningeal involvement
3. Major surgery within 14 days prior to enrollment
4. Peripheral neuropathy (PN)/history of PN ≥ 3
5. Patients who are receiving any other anti-myeloma investigational agents.
6. Patients who receive a live attenuated vaccine within 4 weeks of scheduled study treatment administration.
7. Contraindication to any concomitant medication, including those medications administered for infusion reaction, antiviral, antibacterial, anticoagulation, tumor lysis, or hydration prophylaxis given prior or during to therapy.
8. Patient has any of the following:

   * Human immunodeficiency virus (HIV)-positive with 1 or more of the following:
   * History of acquired immune deficiency syndrome (AIDS)-defining conditions cluster of differentiation 4 (CD4) count <350 cells/mm3
   * Detectable viral load during screening or within 6 months prior to screening
   * Not receiving highly active anti-retroviral therapy
   * Had a change in antiretroviral therapy within 6 months of the start of screening
   * Receiving antiretroviral therapy that may interfere with study treatment as assessed after discussion with the Medical Monitor
   * Hepatitis B infection (ie, hepatitis B surface antigen (HBsAg) or hepatitis B virus (HBV)-DNA positive). Patients with resolved infection (ie, patients who are HBsAg negative but positive for antibodies to hepatitis B core antigen (anti-HBc) and/or antibodies to hepatitis B surface antigen (anti-HBs)) must be screened using real-time polymerase chain reaction (PCR) measurement of HBV DNA levels. Those who are PCR positive will be excluded. In the event the infection status is unclear, quantitative viral levels are necessary to determine the infection status Exception: Participants with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination do not need to be tested for HBV DNA by PCR
   * Active hepatitis C infection as measured by positive Hepatitis C Virus (HCV)-ribonucleic acid (RNA) testing. Participants with a history of HCV antibody positivity must undergo HCV-RNA testing. If a participant with history of chronic hepatitis C infection (defined as both HCV antibody and HCV RNA positive) completed antiviral therapy and has undetectable HCV-RNA 12 weeks following the completion of therapy, the participant is eligible for the study.
   * Chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal. Note that FEV1 testing is required for participants with known or suspected of having COPD or asthma, and participants must be excluded if FEV1 <50% of predicted normal.
   * Moderate or severe persistent asthma within the past 2 years or uncontrolled asthma of any classification. Note that FEV1 testing is required for participants with known or suspected asthma, and participants must be excluded if FEV1 <50% of predicted normal.
   * Severe acute respiratory syndrome (SARS) coronavirus (COV) 2 (SARS-CoV-2) PCR testing is mandated within 5 days prior to enrollment. Exclusion if positive or suspected infection. Also, negative chest imaging needs to be confirmed prior to enrollment.
9. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the experimental agents used in study.
10. Female patient refuses to discontinue breastfeeding her infant during study treatment or within 3 months after receiving the last dose of study treatment.
11. Participant plans to father a child while enrolled in this study or within 3 months after the last dose of study treatment.
12. Presence of the following cardiac conditions:

    * New York Heart Association stage III or IV congestive heart failure
    * Myocardial infarction or coronary artery bypass graft ≤6 months prior to study enrollment
    * History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
    * Uncontrolled cardiac arrhythmia or clinically significant electrocardiogram (ECG) abnormalities
    * Unstable or uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina)
13. Uncontrolled intercurrent illness including but not limited to ongoing or active infection, venous thromboembolic disease, hemorrhage, pulmonary fibrosis, pneumonitis, active autoimmune disease or a documented history of autoimmune disease with the exception of vitiligo, type I diabetes, and prior autoimmune thyroiditis that is currently euthyroid based on clinical symptoms and laboratory testing, or psychiatric illness/social situations within 2 weeks that would limit compliance with study requirements.
14. Active malignancy other than SMM requiring treatment in the past 3 years. Any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, carcinoma in situ, or Stage 0/1 malignancy with minimal risk of recurrence per investigator.
15. Have any condition that, in the opinion of the Investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements. Participants with active, uncontrolled bacterial, fungal, or viral infection, including (but not limited to) HBV, HCV, SARS-CoV-2, and known HIV or AIDS-related illness. Comments regarding specific circumstances follow. Active infection must be resolved at least 21 days prior to enrollment. Patients treated with systemic anti-infective agents within 28 days prior to enrollment are not eligible. Prophylactic use of systemic agents is permitted.
16. Patients with impaired decision-making capacity will not be enrolled on this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease (MRD) (10^-5 sensitivity) | Up to 2 years
  Minimal residual disease (MRD) is defined as 0 residual clonal cells in a bone marrow biopsy sample MRD negativity (10^-5 sensitivity) after 12 cycles, in participants who have been newly diagnosed with Multiple Myeloma receiving Lenalidomide and Low-Dose Dexamethasone (ERd) combination treatment.

SECONDARY OUTCOMES:
Best Overall Response | Up to 24 months
  The best overall response is the best response recorded from the start of the treatment until disease progression (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Will be measured during the first 12 and 24 cycles, in participants who have been newly diagnosed with Multiple Myeloma receiving Lenalidomide and Low-Dose Dexamethasone (ERd) combination treatment.
  Will be measured in months.
Sustained MRD Negativity | Up to 2 years
  The sustained rate of MRD-negativity among participants will be reported. The duration of time in months measured from the first time the participant achieves an MRD-negative bone marrow (BM) biopsy result until the time the participant has relapsed from MRD-negativity objectively documented with an MRD-positive BM result.
Minimal residual disease (MRD) (10^-6 sensitivity) | Up to 2 years
  Minimal residual disease (MRD) negativity ( 10^-6 sensitivity) is defined as 0 residual clonal cells in a bone marrow biopsy anytime in the first 24 cycles, in participants who have been newly diagnosed with Multiple Myeloma receiving Lenalidomide and Low-Dose Dexamethasone (ERd) combination treatment.
Progression-Free Survival (PFS) | Up to 24 months
  Progression-free survival (PFS) among study participants will be assessed during treatment and clinical follow-up. PFS is defined as the time in months from start of treatment until disease progression or death.
Overall Survival | Up to 24 months
  Overall survival (OS) among study participants will be assessed during treatment and clinical follow-up. OS is defined as the time in months from start of treatment until death from any cause.
Incidence of Cytokine Release Syndrome (CRS) | Up to 2 years
  Incidence of cytokine release syndrome (CRS), grade of CRS, and management of potentially recurring CRS. CRS will be evaluated according to the standards released by American Society for Transplantation and Cellular Therapy (ASTCT) criteria in 2019.

CONTACTS AND LOCATIONS:
Overall Officials: Carl O Landgren, MD, Principal Investigator — Professor of Medicine
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No